CLINICAL TRIAL: NCT02477982
Title: Influence of Obesity on Propofol Pharmacokinetics During Cardiac Surgeries Using Cardiopulmonary Bypass: Derivation of a Pharmacokinetic Model
Brief Title: Influence of Obesity on Propofol Pharmacokinetics During Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Ali Ali, Teaching assistant at clinical pharmacy department faculty of pharmacy, Cairo University
Other Study IDs: CL(609)
Record Dates: First submitted 2015-06-14; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
Keywords: Propofol; Cardiopulmonary Bypass; Pharmacokinetics; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- control group: BMI ≤ 25 kgm-2
- obese group: BMI ≥ 30 kgm-2

SUMMARY:
The primary objective of this study is to develop a descriptive and predictive pharmacokinetics model propofol disposition during cardiopulmonary bypass (CPB) in obese and lean patients.

DETAILED DESCRIPTION:
Anaesthesia maintenance upon initiation of CPB will be achieved by propofol (1%) bolus (1 mg/kg TBW) immediately followed by 2 mg/kg TBW/hr infusion that will be continued till weaning from CPB. During CPB an additional propofol bolus doses can be administered to prevent awareness according to the clinical judgment of the responsible anaesthesiologist. Any additional doses given and their timings will be recorded.

Blood samples of 2 ml each will be collected from the arterial line of CPB machine until the end of CPB then from sub-clavin arterial catheter routinely inserted in such surgeries. Sampling process will follow the following schedule; at baseline prior to dosing, followed by samples at 1, 3, 5,7 min after the propofol bolus dose, then every 20 minutes during propofol infusion, just before discontinuation of the propofol infusion and at 1, 3, 5, 7, 10, 20, 30, 60 minutes after the end of infusion. In addition, just before any rescue propofol dose administration, an unscheduled sample will be withdrawn

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 25 kg/m2 or ≥ 30 kg/m2.
* Propofol based maintenance of anaesthesia during CPB.

Exclusion Criteria:

* Pregnant women or lactating mothers.
* Renal (serum creatinine concentration>1.5 or creatinine Cl ≤ 30 ml/min) or hepatic disorders (total bilirubin >1.5 or ≥ 2 fold increase in alanine transferase (ALT) or aspartate transferase (AST).
* Systemic infections.
* Hypoalbuminemia (defined as albumin <3.5 gm/dL).
* Known history of alcohol or drug abuse.
* Administration of aspirin on the day of surgery or warfarin within 7 days preceding surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgery using Cardiopulmonary bypass with moderate hypothermia (defined as core body temperature of 28-32oC).
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Clearance (Cl/) | intraoperative
volume of distribution of first compartment (V1) | intraoperative
Clearance from first to second compartment (Q1) | intraoperative
volume of distribution of second compartment (V1) | intraoperative